CLINICAL TRIAL: NCT03399409
Title: Motivational Interviewing in Physiotherapy for Patients With Low Back Pain: Effects on Adherence to Exercises and on Levels of Incapacity and Pain
Brief Title: Motivational Interviewing in Physiotherapy for Patients With Low Back Pain
Acronym: HELENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HELENA
Record Dates: First submitted 2017-11-29; First posted 2018-01-16 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-11

CONDITIONS: Motivational Interviewing
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing
- Anti-inflammatory information program (Active Comparator)
  Interventions: Behavioral: Anti-inflammatory Information

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivation techniques
  Arms: Motivational Interviewing
Behavioral: Anti-inflammatory Information — Provision of information on anti-inflammatory products
  Arms: Anti-inflammatory information program

SUMMARY:
This study aims to evaluate the efficacy of motivational interviewing (MI) on adherence to exercises and on levels of pain and incapacity in patients who engage in physiotherapy for low back pain. Sixty patients attending a 15-day program of physiotherapy for low back pain were allocated to experimental (EG) and control groups (CG). A regular treatment of physiotherapy with at-home exercises is offered to all participants. On day seven, MI is applied to the EG. The CG receives an anti-inflammatory information program.

ELIGIBILITY:
Inclusion Criteria:

* Adults with low back pain receiving physiotherapy with home exercises

Exclusion Criteria:

* Adults receiving physiotherapy without home exercises or for conditions other than low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in adherence to home exercises | Change from Baseline Performance of Exercises at 2 weeks
  At home exercises checked on the daily Table of Exercises

SECONDARY OUTCOMES:
Change in levels of pain | Change from Baseline Levels of Pain at 2 weeks
  Intensity of pain on the Verbal Pain Intensity Scale. Score range: none, mild, moderate, severe and maximum possible pain
Change in levels of incapacity | Change from Baseline Levels of Incapacity at 2 weeks
  Ability to conduct daily activities on the Roland-Morris Disability Questionnaire. Scores range from 0 to 24, increasing values indicating greater levels of incapacity

CONTACTS AND LOCATIONS:
Overall Officials: Irene P carvalho, Ph.D., Principal Investigator — Universidade do Porto